CLINICAL TRIAL: NCT04608942
Title: Plasma Jet Approach for Refractory Meibomian Gland Dysfunction Patients
Brief Title: Refractory Meibomian Gland Dysfunction and Plasma Jet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Rossen Mihaylov Hazarbassanov, MD, PhD, Associate Professor in Ophthalmology, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31031420.6.0000.5505
Record Dates: First submitted 2020-09-20; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Meibomian Gland Dysfunction; Dry Eye Disease; Evaporative Dry Eye; Inflammation; Tear Film Deficiency
Keywords: meibomian gland dysfunction (MGD); evaporative dry eye disease (E-DED); jett plasma medical lift
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jett Plasma Medical Lift Application (Experimental): In the study group, the plasma jet will be applied to the superior and inferior eyelid margin in both eyes.
  Interventions: Device: Jett Plasma Medical Lift
- Mechanical Debridement (Active Comparator): In the control group, the mechanical debridement of the superior and inferior eyelid margin with a scalpel blade will be performed.
  Interventions: Procedure: Mechanical Debridement

INTERVENTIONS:
Device: Jett Plasma Medical Lift — Plasma Application versus Mechanical Debridement in refractory meibomian gland dysfunction
  Arms: Jett Plasma Medical Lift Application
Procedure: Mechanical Debridement — Plasma Application versus Mechanical Debridement in refractory meibomian gland dysfunction
  Arms: Mechanical Debridement

SUMMARY:
PURPOSE: The investigators propose a new treatment for refractory Meibomian Gland Dysfunction (MGD) patients with plasma jet to remove the hyperkeratinization layer from the lid margin to unblock terminal gland ducts and use thermal stimulation to enhance meibum delivery.

METHODS: A prospective, interventional clinical safety and efficacy trial with 25 patients from the Department of Ophthalmology at Escola Paulista de Medicina (UNIFESP) to determine the efficacy and safety of the treatment of refractory MGD patients with plasma jet on both upper and lower lids. Patients will be submitted to an ophthalmology workup with best-corrected visual acuity (BCVA) (ETDRS chart) and dry eye questionnaires (DEQ-5 and OSDI). Bulbar redness, tear film meniscus height, noninvasive breakup time (NIKBUT), meibography under infrared light will be measured with Keratograph (Oculus®). Following, tear film osmolarity (i-PenTM), meibomian gland expression, and Marx line assessment. All exams were performed at the baseline, 30 days, and 90 days after the plasma jet application.

DETAILED DESCRIPTION:
INTRODUCTION Dry eye disease (DED) is one of the most prevalent conditions at an ophthalmology office that may reach 15 to 40% of prevalence in the population. It is didactically classified as two forms that exist as a continuum: aqueous deficient dry eye (ADDE) and evaporative dry eye (EDE). In EDE patients Meibomian Gland Dysfunction (MGD) is the major etiology in which the insufficient meibum secretion can be decreased by cicatricial (trachoma, ocular pemphigoid, erythema multiforme) and non-cicatricial causes (skin disorders such as acne rosacea and atopic dermatitis, blepharitis).

MGD pathophysiology can be explained by hyposecretion or ducts obstruction, resulting in low delivery of phospholipids and cholesterol that grant stability to the tear film. Hyposecretion of the sebaceous glands can result from intrinsic (age, ethnicity, hormonal profile) and extrinsic factors (chronic blepharitis, Demodex folliculorum infestation, contact lens wear, topical drops). Furthermore, the duct obstruction occurs in a consequence to cicatricial rearrangement of the terminal ducts or by non-cicatricial hyperkeratinization of the lid margins, leading to increased duct pressure, dilatation, and disuse atrophy of the glands.

Questionnaires such as Ocular Surface Disease Index (OSDI) and Dry Eye Questionnaire-5 (DEQ-5) that evaluate the grade of severity of DED and assessment of MGD by noninvasive tear breakup time (BUT) evaluation that measures tear film stability and by meibography under infrared light that analyses gland vitality are central when dealing with any EDE patient.

The treatment of MGD can be very challenging in cases where a clinical approach with non-preserved ocular lubricants, lid hygiene, and warm compresses are not sufficient. Oral tetracyclines can be a good alternative in cases of evident lid inflammation to reduce bacterial colonization and inhibit collagenase action although long-term use intolerance limits its use.

Thermodynamic treatment with a device that performs controlled local heating and massage of the ducts showed clinical improvement and symptoms reduction whereas multiple sessions are necessary. Mechanical debridement of gland ducts terminals with scalpel blade also improved ocular symptoms and gland function of patients with EDE with MGD. A combination of intense pulsed light (IPL) therapy and gland expression has been shown to be an effective treatment to MGD with increases in BUT and improvement of ocular symptoms related to DED.

Plasma jet has been successfully used in Dermatology and is an increasingly popular method for smoothing wrinkles, blunt blepharoplasty, as well as performing thermal ablation for superficial skin layers.

The investigators propose a new treatment for refractory MGD patients with plasma jet with a device used in Dermatology to remove the hyperkeratinization layer from the lid margin to unblock terminal gland ducts and use thermal stimulation to enhance meibum delivery.

METHODS A prospective, interventional clinical safety and efficacy trial to determine the efficacy and safety of the treatment of refractory MGD patients with plasma jet will be conducted at Ophthalmology Department at Escola Paulista de Medicina (UNIFESP) with 25 Caucasian patients.

All patients will be instructed about the study design and will be given full access to the results at any time of the protocol. All will sign an informed consent form and have their identity protected in accordance with patient medical confidentiality. This case series is in accordance with Good Clinical Practices and the Declaration of Helsinki.

Patients will be submitted to an ophthalmology workup with best-corrected visual acuity (BCVA) (ETDRS chart), dry eye questionnaires (DEQ-5 and OSDI), corneal topography, bulbar redness, tear meniscus height, noninvasive breakup time (NBUT), tear film osmolarity, meibography under infrared light, meibomian gland expression and Marx line assessment. All exams will be performed before and 30 days after the plasma jet application.

Patients will be instructed about the procedure by the ophthalmologist and a nurse and the procedure will be performed after topical anesthesia with lidocaine 2.0%. The plasma jet will be applied 3 times on both superior and inferior terminal gland ducts in the lid margins with a 14.4mm tip and intensity of 5 on the device (0,9W) reaching only the superficial epidermis. Patients will receive topical antibiotics and corticosteroids after the procedure. During all periods (90 days) patients will use sodium hyaluronate 0,15% and actinoquinol at the recommended dosage of twice a day.

The software program GraphPad Prism version 7.0 will be used to conduct the statistical analyses. Continuous data distribution will be verified by the Kolmogorov-Smirnov normality test. Data will be analyzed by the Kruskal-Wallis test with the Wilcoxon test considering 2-time points for nonparametric variables and paired t-test for parametric variables. All p values of < 0.05 will indicate statistically significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Refractory meibomian gland dysfunction;
* Previous eyelid hygiene with warm compress in the last 6 months;
* Previous oral intake of antibiotics and antiinflammatories in the last 6 months;
* Previous oral tetracycline treatment for at least one month in the last 6 months;
* DEQ-5 score greater than 6;
* OSDI score greater than 13;
* Tear film osmolarity greater than 308mOsm or a difference between eyes greater than 8 mOsm;
* Meibomian gland expression greater than 8;
* Meibomian gland expression grades 2 or 3 [Nelson 1930];

Exclusion Criteria:

* Cardiac pacemaker or ECG Holter;
* Other electromagnetic device implanted;
* Epilepsy;
* Pregnancy;
* Metal implants in the periocular area;
* Skin diseases in the periocular area;
* Systemic inflammatory diseases;
* Oncological diseases;
* Allergy to local anesthetics;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Dry Eye Questionnaire (DEQ-5) | 30 days
  Dry Eye Questionnaire (DEQ-5) comprises of 5 quick questions and its score ranges from 0 to 22, with lower scores indicating a less severe disease (improvement).
Ocular Surface Disease Index (OSDI) | 30 days
  Ocular Surface Disease Index (OSDI) comprises of 12 questions, each one scored from 0 to 4, and the final score, on a scale from 0 to 100, result from the sum of all values divided by the number of questions answered. Lower scores indicate a less severe disease (improvement).
Bulbar redness | 30 days
  Conjunctival hyperemia will be measured with Keratograph (Oculus®, Inc). This software grades de hyperemia in both nasal and temporal bulbar regions and in the limbal area, with a final score indicating overall ocular surface redness. Greater scores indicate greater hyperemia.
Tear film meniscus height | 30 days
  Tear film meniscus height will be measured with Keratograph (Oculus®, Inc). This software allows individual measurente of the tear film meniscus height (in milimeters) that will be performed in three regions (nasal, central and temporal tear meniscus) and the arithmetic average will be considered to evaluate treatment outcomes, with increased heights indicanting more tear volume.
Non-invasive tear breakup time (NITBUT) | 30 days
  Non-invasive tear breakup time (NITBUT) will be assessed first with Keratograph (Oculus®, Inc). The NITBUT evaluate the tear film stability by registering the time lapse for the first rupture in the tear film to appear. Greater values indicates a more stable tear film.
Tear film osmolarity | 30 days
  Tear film osmolarity will be measured by collecting a micro drop from the tear meniscus with i-Pen (i-Med Pharma, Inc). The tear osmolarity is used to indirect assess occular surface inflammation, with tear osmolalities greater than 308 mOsm or a difference between eyes greater than 8 mOsm indicating tear film disturbance (Dry Eye WorkShop II - DEWS II 2017).
Meibomian gland expression | 30 days
  Meibomian gland expression will be performed using Meibomian Gland Evaluator (MGE), a special devide with precise pression, that will allow to assess meibomian glands in the slit lamp. This devices acts on five glands at a time, so meibum deliverance can be judged in quantity (is there any gland duct obstructed?) and quality (is meibum clear, cloudy or opaque?).

SECONDARY OUTCOMES:
Dry Eye Questionnaire (DEQ-5) | 90 days
  Dry Eye Questionnaire (DEQ-5) comprises of 5 quick questions and its score ranges from 0 to 22, with lower scores indicating a less severe disease (improvement).
Ocular Surface Disease Index (OSDI) | 90 days
  Ocular Surface Disease Index (OSDI) comprises of 12 questions, each one scored from 0 to 4, and the final score, on a scale from 0 to 100, result from the sum of all values divided by the number of questions answered. Lower scores indicate a less severe disease (improvement).
Bulbar redness | 90 days
  Conjunctival hyperemia will be measured with Keratograph (Oculus®, Inc). This software grades de hyperemia in both nasal and temporal bulbar regions and in the limbal area, with a final score indicating overall ocular surface redness. Greater scores indicate greater hyperemia.
Tear film meniscus height | 90 days
  Tear film meniscus height will be measured with Keratograph (Oculus®, Inc). This software allows individual measurente of the tear film meniscus height (in milimeters) that will be performed in three regions (nasal, central and temporal tear meniscus) and the arithmetic average will be considered to evaluate treatment outcomes, with increased heights indicanting more tear volume.
Non-invasive tear breakup time (NITBUT) | 90 days
  Non-invasive tear breakup time (NITBUT) will be assessed first with Keratograph (Oculus®, Inc) and then with florescein dye. The NITBUT evaluate the tear film stability by registering the time lapse for the first rupture in the tear film to appear. Greater values indicates a more stable tear film.
Tear film osmolarity | 90 days
  Tear film osmolarity will be measured by collecting a micro drop from the tear meniscus with i-Pen (i-Med Pharma, Inc). The tear osmolarity is used to indirect assess occular surface inflammation, with tear osmolalities greater than 308 mOsm or a difference between eyes greater than 8 mOsm indicating tear film disturbance (Dry Eye WorkShop II - DEWS II 2017).
Meibomian gland expression | 90 days
  Meibomian gland expression will be performed using Meibomian Gland Evaluator (MGE), a special devide with precise pression, that will allow to assess meibomian glands in the slit lamp. This devices acts on five glands at a time, so meibum deliverance can be judged in quantity (is there any gland duct obstructed?) and quality (is meibum clear, cloudy or opaque?).

CONTACTS AND LOCATIONS:
Overall Officials: Rossen M Hazarbassanov, MD PhD, Principal Investigator — Associate Professor in Ophthalmology (Federal University of Sao Paulo - UNIFESP)
Locations (2):
- Brazil (2):
  - Departamento de Oftalmologia da Escola Paulista de Medicina - UNIFESP, São Paulo, São Paulo
  - Department of Ophthalmology, UNIFESP&EPM, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Nichols KK, Foulks GN, Bron AJ, Glasgow BJ, Dogru M, Tsubota K, Lemp MA, Sullivan DA. The international workshop on meibomian gland dysfunction: executive summary. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1922-9. doi: 10.1167/iovs.10-6997a. No abstract available. PMID 21450913
- [Background] Scott E Schachter, Aubrey Schachter, Milton M Hom, Scott G Hauswirth; Prevalence of MGD, blepharitis, and demodex in an optometric practice.. Invest. Ophthalmol. Vis. Sci. 2014;55(13):49.
- [Background] Stapleton F, Alves M, Bunya VY, Jalbert I, Lekhanont K, Malet F, Na KS, Schaumberg D, Uchino M, Vehof J, Viso E, Vitale S, Jones L. TFOS DEWS II Epidemiology Report. Ocul Surf. 2017 Jul;15(3):334-365. doi: 10.1016/j.jtos.2017.05.003. Epub 2017 Jul 20. PMID 28736337
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Chalmers RL, Begley CG, Caffery B. Validation of the 5-Item Dry Eye Questionnaire (DEQ-5): Discrimination across self-assessed severity and aqueous tear deficient dry eye diagnoses. Cont Lens Anterior Eye. 2010 Apr;33(2):55-60. doi: 10.1016/j.clae.2009.12.010. Epub 2010 Jan 25. PMID 20093066
- [Background] Tian L, Qu JH, Zhang XY, Sun XG. Repeatability and Reproducibility of Noninvasive Keratograph 5M Measurements in Patients with Dry Eye Disease. J Ophthalmol. 2016;2016:8013621. doi: 10.1155/2016/8013621. Epub 2016 Apr 12. PMID 27190639
- [Background] Olson MC, Korb DR, Greiner JV. Increase in tear film lipid layer thickness following treatment with warm compresses in patients with meibomian gland dysfunction. Eye Contact Lens. 2003 Apr;29(2):96-9. doi: 10.1097/01.ICL.0000060998.20142.8D. PMID 12695712
- [Background] Dougherty JM, McCulley JP, Silvany RE, Meyer DR. The role of tetracycline in chronic blepharitis. Inhibition of lipase production in staphylococci. Invest Ophthalmol Vis Sci. 1991 Oct;32(11):2970-5. PMID 1917401
- [Background] Korb DR, Blackie CA. Restoration of meibomian gland functionality with novel thermodynamic treatment device-a case report. Cornea. 2010 Aug;29(8):930-3. doi: 10.1097/ICO.0b013e3181ca36d6. PMID 20531168
- [Background] Korb DR, Blackie CA. Debridement-scaling: a new procedure that increases Meibomian gland function and reduces dry eye symptoms. Cornea. 2013 Dec;32(12):1554-7. doi: 10.1097/ICO.0b013e3182a73843. PMID 24145633
- [Background] Arita R, Mizoguchi T, Fukuoka S, Morishige N. Multicenter Study of Intense Pulsed Light Therapy for Patients With Refractory Meibomian Gland Dysfunction. Cornea. 2019 Feb;38(2):e4. doi: 10.1097/ICO.0000000000001779. No abstract available. PMID 30418276
- [Background] Tremblay JF, Moy R. Treatment of post-auricular skin using a novel plasma resurfacing system: an in vivo clinical and histologic study (abstract). Lasers Surg Med. 2004;34 (suppl 16):25.
- [Background] Vanden Bosch ME, Wall M. Visual acuity scored by the letter-by-letter or probit methods has lower retest variability than the line assignment method. Eye (Lond). 1997;11 ( Pt 3):411-7. doi: 10.1038/eye.1997.87. PMID 9373488
- [Background] Marx E. Uber vitale farbungen am auge und an den lidern. I. Uber anatomie, physiologie und pathologie des Aagenlidrandes und der tranenpunkte. Graefes Arch Clin Exp Ophthalmol. 1924;114:465-82.